CLINICAL TRIAL: NCT05106465
Title: Konect-MF: A Study to Explore Association Patterns Between Digital Outcome Assessments From the Konectom™ Platform and MRI Measures of Brain Tissue Damage
Brief Title: A Study to Explore Association Patterns Between Digital Outcome Assessments From the Konectom™ Platform and Magnetic Resonance Imaging (MRI) Measures of Brain Tissue Damage
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 888MS008
Record Dates: First submitted 2021-10-20; First posted 2021-11-03 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis (MS)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Konectom: Participants with a diagnosis of MS or clinically isolated syndrome who are enrolled in Multiple Sclerosis Partners Advancing Technology and Health Solutions (MS PATHS) and who own a smartphone model compatible with the Konectom platform will be enrolled.
  Interventions: Device: Konectom platform

INTERVENTIONS:
Device: Konectom platform — Administered as specified in the treatment arm.

SUMMARY:
The purpose of the study is to explore association patterns between digital outcome assessments from Konectom and MRI measures of brain tissue damage.

ELIGIBILITY:
Inclusion Criteria:

* Should be enrolled in multiple sclerosis partners advancing technology and health solutions (MS PATHS).
* Participant (or participant's legal representative) has the ability to understand the purpose and risks of the study, to provide signed and dated informed consent, and to authorize the use of confidential health information in accordance with national and local privacy regulations.
* Should have literacy of written language in which the software and Instructions for use are displayed (User Interface [UI], Instructions).

Exclusion Criteria:

* Unable or unwilling to provide informed consent.
* Inability to use a smartphone as per physician's opinion.
* Not owning a Konectom-compatible smartphone.
* Other unspecified reasons that, in the opinion of the Investigator or Biogen, make the participant unsuitable for participation in the sub-study. A participant only needs to complete the assessments deemed necessary by the Investigator.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes participants with a diagnosis of MS who are enrolled in MS PATHS.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Correlation Between Konectom Tests and MRI Measures of Brain Tissue Damage | Up to 1 year
  Konectom tests include cognitive processing speed test (CPST), pinching test, drawing test, static balance test (SBT)/u-turn test (UTT) and 6-minute walking test (6MWT).

SECONDARY OUTCOMES:
Correlation Between Konectom Tests and Deep Radiomic Feature Set Extracted From Fluid-attenuated Inversion Recovery (FLAIR) Hyperintense MS Lesions Using 3D-T1 and 3D FLAIR Data | Up to 1 year
  Konectom tests include CPST, pinching test, drawing test, SBT/UTT and 6MWT.
Correlation Between Konectom Tests and Deep Radiomic Feature Set Extracted From the Normal Appearing White Matter Using 3D-T1 and 3D FLAIR Data | Up to 1 year
  Konectom tests include CPST, pinching test, drawing test, SBT/UTT and 6MWT.
Correlation Between Konectom Tests and Deep Radiomic Feature Set Extracted From the Cortex Using 3D-T1 and 3D FLAIR Data | Up to 1 year
  Konectom tests include CPST, pinching test, drawing test, SBT/UTT and 6MWT.
Correlation Between Konectom Tests and Deep Radiomic Feature Set Extracted From Deep Grey Matter Using 3D-T1 and 3D FLAIR Data | Up to 1 year
  Konectom tests include CPST, pinching test, drawing test, SBT/UTT and 6MWT.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Multiple Sclerosis Centre, Dresden, Germany

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/